CLINICAL TRIAL: NCT06063850
Title: A Multi-center, Phase 1/2a, First-in-human (FIH) Study Investigating the Safety, Tolerability, and Efficacy of AMT-260 in Adults With Unilateral Refractory Mesial Temporal Lobe Epilepsy (MTLE) Administered Via Magnetic Resonance Imaging (MRI)-Guided Convection-enhanced Delivery (CED)
Brief Title: AMT-260 Gene Therapy Study in Adults With Unilateral Refractory Mesial Temporal Lobe Epilepsy
Acronym: GenTLE
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: UniQure Biopharma B.V. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CT-AMT-260-01
Record Dates: First submitted 2023-09-01; First posted 2023-10-03 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Mesial Temporal Lobe Epilepsy
Keywords: Epilepsy; Temporal Lobe; Hippocampal Sclerosis; Epileptic Syndromes
MeSH Terms: conditions — Epilepsy; Hippocampal Sclerosis; Epileptic Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- AMT-260 (Experimental): Cohort 1: AMT-260 starting dose (1.0x 10E12 gc/mL). Cohort 2: AMT-260 adapted dose (6.0x 10E11 gc/mL or 3.0x 10E12 gc/mL).
  Interventions: Genetic: AAV9-hSyn1-miGRIK2

INTERVENTIONS:
Genetic: AAV9-hSyn1-miGRIK2 — AMT-260 is an AAV9 gene therapy product that locally delivers miRNA silencing technology to target the GRIK2 gene and suppress aberrantly expressed GluK2 containing kainate receptors. Intervention will be a one-time intracerebral administration of AMT-260.
  Other Names: AMT-260

SUMMARY:
The main goals of this clinical study are to learn if AMT-260 is safe and tolerable and works to reduce the frequency of seizures in adults with unilateral mesial temporal lobe epilepsy (MTLE).

DETAILED DESCRIPTION:
In this first clinical study of AMT-260, two dose levels will be studied to find the best dose of AMT-260. All eligible participants will receive AMT-260 at one of the two dose levels (i.e., there is no placebo in this study).

AMT-260 is intended for a one-time administration, without the need to remove or destroy any part of the brain. Participation in this study would not prevent later pursuit of other treatment options.

Participants will be monitored through study site visits, telephone calls, blood tests, and questionnaires about how their seizures affect daily life. Participants will record seizures using an electronic seizure diary.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of unilateral refractory MTLE
* History of seizures with an average of ≥ 2 documented focal impaired awareness seizures or focal to bilateral tonic-clonic seizures per 30-day period in the 3 months prior to screening.
* On a stable type and dose regimen of up to a maximum of 4 approved Anti Seizure Drugs for at least 6 months prior to screening.
* Confirmed unilateral hippocampal pathology and concordant unilateral seizure focus
* No evidence of focal neurocognitive dysfunction, inconsistent with disease pathology- related MRI and/or (18F)FDG-PET findings.
* Women of childbearing potential (WOCBP) and fertile male subjects must be willing and able to use highly effective methods of birth control consistently and correctly throughout the study.
* For WOCBP only: Negative pregnancy test.

Exclusion Criteria:

* Implanted devices that would contraindicate MRI; MRI-compatible devices must be implanted ≥3 months prior to Screening (vagus nerve stimulation devices will be up to discretion of the Investigator).
* Any other contraindications for generalized anesthesia or surgery.
* Medications that could confound clinical (e.g., antipsychotic medication and anti-viral therapy) and laboratory evaluations or could affect a participant's safety or their ability to undergo the neurosurgical procedure or comply with the procedures and study visit schedule.
* Any seizures with contralateral or extra-temporal icta onset captured on EEG.
* Dementia or other progressive neurological disorders and progressive brain lesions.
* Previous major disease-unrelated neurosurgical intervention due to intracranial tumor, trauma, or bleeding and/or history of previous intracranial surgery for treatment of epileptic seizures, not including diagnostic stereo-EEG.
* Magnetic resonance imaging evidence of epileptogenic, extra-temporal lesions, or dual temporal lobe pathology.
* Inadequate vaccination status (including flu shots and other relevant immunizations such as COVID-19 per local guidelines and regulations).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-06-12 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2031-12 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of AMT-260 in adults with unilateral refractory MTLE. | 1 year
  Occurrence of Adverse Events during the period of 1 year after AMT-260 administration, including seriousness, severity, and causal relationship to AMT-260.

SECONDARY OUTCOMES:
To evaluate first signs of efficacy of AMT-260. | 1 year
  Change in seizure frequency, comparing baseline to the 1 year period after AMT-260 administration.
To evaluate the biodistribution properties of AMT-260. | 1 year
  Blood, urine, saliva, and CSF samples will be collected and evaluated for vector DNA shedding at each timepoint.

OTHER OUTCOMES:
To evaluate the long-term safety and efficacy of AMT-260 in adults with unilateral refractory MTLE. | up to 5 years
  Occurrence of Adverse Events during the period of 1 to 5 years after AMT-260 administration, including seriousness.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Lead, Study Director — uniQure France SAS
Locations (18):
- United States (18):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Mayo Clinic Arizona, Phoenix, Arizona
  - Stanford University, Palo Alto, California
  - Mayo Clinic Florida, Jacksonville, Florida
  - Kansas University Medical Center, Kansas City, Kansas
  - Johns Hopkins School of Medicine, Baltimore, Maryland
  - Midatlantic Epilepsy and Sleep Center, Bethesda, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Corewell Health, Grand Rapids, Michigan
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Northeast Regional Epilepsy Group, Hackensack, New Jersey
  - Robert Wood Johnson Hospital, New Brunswick, New Jersey
  - Cleveland Clinic, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Allegheny Health Network, Pittsburgh, Pennsylvania
  - Baylor Scott & White Medical Center, Austin, Texas
  - Medical College of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- See also: : Sponsor web page about this Phase 1/2a clinical study of AMT-260 — https://www.uniqure.com/programs-pipeline/phase-i-iia-clinical-trial-of-amt-260